CLINICAL TRIAL: NCT03384823
Title: A Randomized, Double-Blind, Placebo-Controlled, First-In-Human Study of Orally Administered EDP-938 to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses (SAD), Multiple Ascending Doses (MAD) and the Effect of Food on EDP-938 Pharmacokinetics in Healthy Subjects
Brief Title: A Study of EDP-938 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Collaborators: Pharmaceutical Research Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EDP-938-001
Record Dates: First submitted 2017-12-20; First posted 2017-12-27 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: RSV Infection
Keywords: First-in-Human; Single Ascending Dose; Multiple Ascending Dose
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — EDP-938

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- EDP-938 SAD Cohorts (Experimental): EDP-938 Dose 1, Dose 2, Dose 3, Dose 4, Dose 5, and Dose 6 oral suspension, once daily in one single administration
  Interventions: Drug: EDP-938
- EDP-938 MAD Cohorts (Experimental): EDP-938 Dose 1, Dose 2, Dose 3, and Dose 4 oral suspension, once daily for 7 days
  Interventions: Drug: EDP-938
- EDP-938 SAD Placebo Cohort (Placebo Comparator): Matching placebo, oral suspension, once daily in one single administration
  Interventions: Drug: Placebo
- EDP-938 MAD Placebo Cohort (Placebo Comparator): Matching placebo, oral suspension, once daily for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EDP-938 — Subjects will receive either a single dose of EDP-938 on Day 1 only (SAD) or a single dose of EDP-938 starting on Day 1 through Day 7 (MAD).
  Arms: EDP-938 MAD Cohorts; EDP-938 SAD Cohorts
Drug: Placebo — placebo to match EDP-938
  Arms: EDP-938 MAD Placebo Cohort; EDP-938 SAD Placebo Cohort

SUMMARY:
This randomized, double-blind, placebo-controlled study will assess the safety, tolerability, and pharmacokinetics of single and multiple orally administered doses of EDP-938 in healthy adult subjects

DETAILED DESCRIPTION:
The first phase assesses single ascending doses for EDP-938 (active drug or placebo) in healthy subjects. A "fasted" and "fed" two-part cohort will also assess food effect.

The second phase assesses multiple ascending doses (active drug or placebo) for 7-days in healthy subjects.

Each cohort within each phase will enroll a total of 8 subjects who will be randomized to receive EDP-938 or placebo. The cohort assessing food effect will enroll 10 subjects randomized to receive EDP-938 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* An informed consent document signed and dated by the subject.
* Healthy male and female subjects of any ethnic origin between the ages of 18 and 55 years, inclusive.

Exclusion Criteria:

* Clinically relevant evidence or history of illness or disease.
* Pregnant or nursing females.
* History of febrile illness within 7 days prior to the first dose of study drug or subjects with evidence of active infection.
* A positive urine drug screen at screening or Day -1.
* Current tobacco smokers or use of tobacco within 3 months prior to screening.
* Any condition possibly affecting drug absorption (e.g., gastrectomy, cholecystectomy).
* History of regular alcohol consumption.
* Participation in a clinical trial within 30 days prior to the first dose of study drug.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2018-07-03 (Actual)

PRIMARY OUTCOMES:
Safety measured by adverse events, physical exams, vital signs, 12-lead electrocardiograms (ECGs) and clinical lab results (including chemistry, hematology, and urinalysis). | Up to 8 days

SECONDARY OUTCOMES:
Cmax of EDP-938 | Up to 5 Days
Cmax of EDP-938 | Up to 11 Days
AUC of EDP-938 | Up to 5 Days
AUC of EDP-938 | Up to 11 Days

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Inc, Study Director — Enanta Pharmaceuticals, Inc
Locations (1):
- Pharmaceutical Research Associates, Inc.,, Lenexa, Kansas, United States